CLINICAL TRIAL: NCT07133425
Title: A Phase 2 Platform Study of Immunomodulatory Compounds in ICI-refractory Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1996; NCI-2025-06144 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-08-19; First posted 2025-08-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer; ICI-refractory
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase II biomarker study of SAR445877 (Experimental): Will receive SAR445877 by vein over about 60 minutes every 2 weeks, on Day 1 of each 14-day cycle.
  Interventions: Drug: SAR445877

INTERVENTIONS:
Drug: SAR445877 — Given by IV

SUMMARY:
To learn if SAR445877 can help to control locally advanced or metastatic NSCLC in patients who have previously received ICI therapy.

DETAILED DESCRIPTION:
Primary Objectives

* To identify early efficacy signals for SAR445877 in ICI-exposed NSCLC participants
* Identify biomarkers related to the mechanism of action in SAR445877 and predictive of response/resistance in ICI-exposed NSCLC participants

ELIGIBILITY:
Eligibility Criteria

1. Ability to understand and willingness to sign informed consent form (ICF) prior to initiation of the study and any study procedures.
2. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of SAR445877 in participants <18 years of age, children are excluded from this study.
3. Participants with histologically documented locally advanced or metastatic NSCLC who have had disease progression after treatment with all available therapies for metastatic disease that are known to confer clinical benefit, or are intolerant to treatment, or refuse standard treatment:
4. Prior immune checkpoint inhibitor (anti-PD-(L)1) exposure. Participants need to have received at least 6 weeks of exposure to anti-PD-(L)1 and developed disease progression. Treatment with neoadjuvant or adjuvant ICI is acceptable if participant developed progression within one year of start of ICI therapy.
5. One lesion suitable for repeat biopsy without significant risk to the participant.
6. Measurable disease per RECIST v1.1.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 .
8. Adequate organ and marrow function as defined below, obtained before study treatment initiation:

   1. Hemoglobin >9.0 g/dL
   2. Absolute neutrophil count ≥1000/mcL
   3. Platelets ≥75,000/mcL
   4. Total bilirubin ≤1.5 institutional upper limit of normal (ULN). Documented Gilbert syndrome is allowed if total bilirubin is ≤3 × ULN.
   5. AST/ALT ≤2.5 × institutional ULN. Transaminases up to 5 × ULN in the presence of liver metastases.
   6. Measured or calculated creatinine clearance (CrCl; glomerular filtration rate can also be used in place of creatinine or CrCl) ≥30 mL/min (CrCl should be calculated per institutional standard).
   7. For participants not receiving therapeutic anticoagulation: international normalized ratio or activated partial thromboplastin time ≤1.5 × ULN. For participants receiving therapeutic anticoagulation: stable anticoagulant regimen.
9. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test result at screening.
10. WOCBP must agree to use highly effective contraception for the duration of study participation and for 60 days after completion of study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a post-menopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this study must also agree to use adequate contraception for the duration of study participation and for 60 days after completion of study treatment. In addition, male participants must be willing to refrain from sperm donation during this time.
11. Willing to undergo mandatory biopsies and blood collections as required by the study.
12. Participants with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and participant is clinically stable without requirement of steroid treatment for ≥ 7 days prior to the first dose of study treatment.
13. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

Exclusion Criteria

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs.
2. Participants who are pregnant or breastfeeding.
3. Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Participants with a condition requiring systemic treatment with either corticosteroid (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study treatment initiation. Inhaled or topical steroids, and adrenal replacement steroid doses, are permitted in the absence of active autoimmune disease.
5. History of interstitial lung disease (ILD) or checkpoint inhibitor-induced pneumonitis.
6. Known history of positive test for human immunodeficiency virus or known acquired immunodeficiency syndrome.
7. Acute or chronic hepatitis B virus or hepatitis C virus infection. Prior viral exposure with cleared or fully treated infection based on negative HCV viral load is permitted.
8. Previous solid organ or allogeneic hematopoietic stem cell transplant.
9. Active infection requiring IV antibiotics or other uncontrolled intercurrent illness requiring hospitalization.
10. Significant cardiovascular/cerebrovascular disease, including stroke, myocardial infarction, or prolonged QTc (> 480msec) within 3 months. Participants on beta blockers must be able to stop beta blockers for duration of their time on study treatment period when applicable.
11. Participants who have not recovered from AEs due to prior anticancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia, hearing loss, grade 2 neuropathy or endocrinopathy managed with hormone replacement therapy.
12. Participants who have previously been treated with PD-1, PD-L1, or CTLA-4 inhibitors and required permanent discontinuation or systemic immunosuppression (e.g. immune inhibitory monoclonal antibodies) due to irAEs.
13. Participants who are receiving any other investigational agents.
14. Treatment with a live, attenuated vaccine within 4 weeks prior to study treatment initiation, or anticipation of need for such a vaccine during the course of the study or within 5 months after the last dose of study treatment. Non-live COVID vaccines will be allowed on study, but it is recommended to avoid their use during the first treatment cycle (from 3 days prior to Cycle 1 Day 1 through Cycle 2 Day 3).
15. Participants must have adequate washout from prior therapy at the time of study treatment initiation: 4 weeks from major surgery; 4 weeks from antibody-based therapy; 3 weeks from prior PD-(L)1 inhibitor exposure; 2 weeks or 5 half-lives (whichever is shorter) from any targeted therapy or small molecule therapy; 3 weeks or 5 half-lives (whichever is shorter) from chemotherapy or 6 weeks in the case of certain therapies (e.g., extensive radiotherapy, mitomycin C, and nitrosoureas); and 2 weeks from radiation therapy. Palliative radiotherapy is permitted for a preexisting lesion, provided it does not interfere with the assessment of tumor target lesions (e.g., the lesion to be irradiated must not be a site of measurable disease).
16. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, ductal carcinoma in situ, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
17. Has a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the study.
18. Inability to comply with the study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Vokes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org